CLINICAL TRIAL: NCT06451276
Title: The Effectiveness of Adhesive Versus Conventional Nasoalveolar Molding on Alveolar Ridge, Nasal and Labial Growths in Children With Unilateral Cleft Lip and Palate
Brief Title: The Effectiveness of Adhesive Versus Conventional Nasoalveolar Molding on Children With Unilateral Cleft Lip and Palate
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Farghly Abdelnaeem Ahmed, Doctor, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NAM in unilateral cleft
Record Dates: First submitted 2024-05-31; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Cleft Lip and Palate
MeSH Terms: conditions — Cleft Lip | interventions — Nasoalveolar Molding

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Adhesive nasoalveolar molding (GS-NAM) (Active Comparator): 3D (3 dimensional ) printed conventional NAM in thickness of 2 mm. The cleft area will be blocked in software, and NAM will be fabricated using a 3D (3 dimensional ) printer. Soft acrylic resin will be added to make pressure area and reduction in opposing for relief. The appliance will be evaluated and adjusted monthly. A nasal stent will be fabricated when the cleft is 5mm
  Interventions: Device: Nasoalveolar molding in unilateral cleft lip and palate
- Conventional nasoalveolar molding (Experimental): (positive control group) comprises 10 cases of unilateral cleft lip and palate that will be scheduled for construction of 3D (3 dimensional ) printed conventional NAM in thickness of 2 mm. The cleft area will be blocked in software, and NAM will be fabricated using a 3D printer. Soft acrylic resin will be added to make pressure area and reduction in opposing for relief. The appliance will be evaluated and adjusted monthly. A nasal stent will be fabricated when the cleft is 5mm
  Interventions: Device: Nasoalveolar molding in unilateral cleft lip and palate
- normal children (No Intervention): normal children which will be compared with groups 1 and 2 for results evaluation

INTERVENTIONS:
Device: Nasoalveolar molding in unilateral cleft lip and palate — compare the effectiveness of adhesive nasoalveolar molding (GS-NAM) and conventional nasoalveolar molding on the alveolar ridge, nasal, and labial growth in children with unilateral cleft lip and palate
  Other Names: NAM
  Arms: Adhesive nasoalveolar molding (GS-NAM); Conventional nasoalveolar molding

SUMMARY:
The present study will compare the effectiveness of adhesive nasoalveolar molding (GS-NAM) and conventional nasoalveolar molding on the alveolar ridge, nasal, and labial growth in children with unilateral cleft lip and palate.

objectives: -

1. Evaluation of the anatomical position of the greater and lesser segments of the maxilla related to a stable midline anatomical point.
2. Evaluation of the nasal symmetry.

DETAILED DESCRIPTION:
cleft lip and palate can manifest as an independent anomaly, be associated with a syndrome, or present as a complex condition. Unilateral clefts are notably more common, occurring nine times more frequently than bilateral clefts. Additionally, it predominantly affects males, with a male-to-female ratio of 2:1. Common clinical features in unilateral cleft lip and palate cases involve structural changes in the nose, lip, palate, and alveolar arch. Peri-oral tissues lack continuity, and on the affected side of the nose, you can observe wider nostrils and a downward-pointing alar rim. Additionally, the columella and nasal tip shift towards the unaffected or normal side, accompanied by the displacement of the maxillary alveolar segments towards the lateral side.

Conventional treatment for cleft lip and palate historically comprised numerous surgical procedures, including secondary revisions and alveolar bone grafting. However, even with these multiple interventions, concerns persisted regarding suboptimal aesthetics. Therefore, the pursuit of non-surgical treatment options that can mitigate the severity of this deformity during early life is greatly desirable. The introduction of the presurgical Nasoalveolar molding (NAM) procedure has offered an alternative, allowing for the avoidance of traditional secondary surgeries while achieving improved outcomes. . These interventions should be initiated within the narrow time frame from birth to four months, as estrogen levels decrease within the first four months after birth, making this period optimal for tissue manipulation.

ELIGIBILITY:
Inclusion Criteria:

* Age: 1- 8 weeks.
* Gender: male and female.
* Patients with a unilateral cleft alveolus and lip.
* No developmental syndromes or atypical cleft pathology in medical history.
* No previous history of unilateral CLP correction.
* Motivated parents toward the treatment.

Exclusion Criteria:

* Patients with a bilateral cleft alveolus and lip
* Syndromic patient
* Uncooperative caregiver

Ages: 7 Days to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-07-20 (Estimated); Primary Completion 2025-07-20 (Estimated); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
Posterior ends of alveolar crest | 3 months
  width between the most posterior ends of the alveolar crest in the greater segment and lesser segment
Middle ends of alveolar crest | 3 months
  width between the middle parts of the cleft palate (The intersection points between the palatally extended buccal frenum sulcus line and the palatal gingival groove in the greater and lesser segment
Anterior ends of alveolar crest | 3 months
  The widths of the cleft gap (The anterior endpoint of the alveolar crest in the greater and lesser segment)
Mid line of maxilla | 3 months
  Inc-Sagittal: - Perpendicular distance from Inc point (The intersection points between the labial frenum-incisive papilla point line and the alveolar crest of the premaxilla in the greater segment) to sagittal line (The perpendicular line to the PG-PL line)
Angulation of maxilla | 3 months
  Mid-Inc)-Sagittal: - Angle among Inc point, midpoint in PG -PL, and sagittal line

SECONDARY OUTCOMES:
Alar base width | 3 months
  Total width correction of alar base width.
Columella length. | 3 months
  Columella length correction
Columella angle deviation. | 3 months
  Columella angle deviation correction
Nostril height and width on the cleft side. | 3 months
  Nostril height and width on the cleft side correction
Nostril height and width on the non-cleft side | 3 months
  Nostril height and width on the non-cleft side correction
Nasal ridge deviation. | 3 months
  Nasal ridge deviation correction

CONTACTS AND LOCATIONS:
Overall Officials: Adel F Hassan, Phd, Study Director — Fucalty of dental medicine
Locations (2):
- Egypt (2):
  - Faculty of dental medicine, Cairo
  - Faculty of Dental Medicine (Boys, Cairo), Al- Azhar University, Cairo

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: 4 months
Access Criteria: all IPD that underlie results in a publication
URL: http://Ahmedfarghly0@gmail.com